CLINICAL TRIAL: NCT01340430
Title: Neoadjuvant Therapy With FEC Followed by Weekly Paclitaxel and Concurrent Trastuzumab in Her2 Positive Non Operable Breast Cancer. Phase II Study.
Brief Title: Neoadjuvant 5-fluorouracil, Epirubicin and Cyclophosphamide (FEC) Followed by Weekly Paclitaxel and Trastuzumab in Her2 Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lucia Del Mastro,MD (Other)
Responsible Party: Sponsor-Investigator, Lucia Del Mastro,MD, md, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Organization: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEOHER-021; 2010-021600-24 (EudraCT Number)
Record Dates: First submitted 2011-04-06; First posted 2011-04-22 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: HER-2 Positive Breast Cancer
Keywords: her2 positive breast cancer; her2 positive non operable breast cancer; her2 positive locally advanced breast cancer; neoadjuvant trastuzumab; pathologic complete response
MeSH Terms: conditions — Pathologic Complete Response | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FEC-paclitaxel-trastuzumab (Experimental): fluorouracil 600 mg/m2; epirubicin 90 mg/m2; cyclophosphamide 600 mg/m2 for 4 cycles followed by paclitaxel 80 mg/m2/week in combination with trastuzumab for 12 weeks
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — neoadjuvant FEC (fluorouracil, epirubicin, cyclophosphamide) followed by weekly paclitaxel and concomitant trastuzumab
  Other Names: herceptin

SUMMARY:
The main purpose of this study is to confirm the high pathologic complete response rate after neoadjuvant chemotherapy with FEC followed by weekly paclitaxel and concurrent trastuzumab in Human Epidermal growth factor receptor2 (HER2) positive non operable breast cancer

ELIGIBILITY:
Inclusion Criteria

1. Performance StatusEstearn Cooperative Oncology Group (ECOG) 0-1
2. Histologically confirmed invasive breast cancer,
3. Primary tumour greater ≥ 2 cm diameter, measured by clinical examination and mammography or echography or Nuclear Magnetic Resonance (NMR) candidate to neoadjuvant chemotherapy ,
4. Any N,
5. No evidence of metastasis (M0);
6. Over expression and/or amplification of HER2 in the invasive component of the primary tumour according to one of the following definitions:
7. 3+ over expression by immunohistochemistry (IHC) (> 30% of invasive tumour cells),
8. 2+ or 3+ (in 30% o less neoplastic cells) overexpression by IHC and in situ hybridization (FISH/CISH) test demonstrating Her2 gene amplication ,
9. Her 2 gene amplication by FISH/CISH (ratio > 2.2);
10. Known hormone receptor status
11. Hematopoietic status:

    1. absolute neutrophil count ≥ 1.5 x 109/L,
    2. platelet count ≥ 100 x 109/L,
12. Hepatic status:

    1. serum total bilirubin ≤ 1.5 x ULN. In the case of known Gilbert's syndrome a higher serum total bilirubin (< 2 x ULN) is allowed,
    2. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN,
    3. alkaline phosphatase ≤ 2.5 times ULN;
13. Renal status:

    a. Creatinine ≤ 2.0 mg/dL;
14. Cardiovascular:

    a. baseline left ventricular ejection fraction (LVEF) ≥ 50% measured by echocardiography or multigate acquisition scan (MUGA);
15. For women of childbearing potential negative serum pregnancy test
16. Written informed consent.

Exclusion Criteria:

1. Male gender
2. Pregnant or lactating women
3. Received any prior treatment for primary invasive breast cancer
4. Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension (> 180/110), unstable diabetes mellitus, dyspnoea at rest or chronic therapy with oxygen;
5. Active or uncontrolled infection,
6. Dementia altered mental status or any psychiatric condition that would prevent the under standing or rendering of informed consent,
7. Concurrent neoadjuvant cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy other than the trial therapies),
8. Previous or concomitant malignancy within the past 3 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix.
9. Concurrent disease or condition that would have make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-03; Primary Completion 2015-12 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
pathologic complete response | at definitive surgery within 4 weeks after the last dose of paclitaxel and concurrent trastuzumab

SECONDARY OUTCOMES:
safety and tolerability | one year
  safety and tolerability will be assessed by standard clinical and laboratory tests (hematology, serum chemistry). Toxicity grade is defined by the NCI Common Toxicity Criteria (CTC) Adverse Event (AE) v 3.0
cardiotoxicity | one year
disease free survival | one year
overall survival | one year
rate of conversion from radical to conservative surgery | definitive surgery
potential biomarkers of trastuzumab resistance | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Del Mastro, MD, Principal Investigator — National Institute For Cancer Reasearch
Locations (6):
- Italy (6):
  - Istituto Nazionale per La Ricerca sul Cancro (IST), Genoa, Ge
  - Ospedale S. Maria della Misericordia - Oncologia Medica, Perugia, PG
  - Fondazione del Piemonte per l'Oncologia - IRCC di Candiolo, Candiolo, TO
  - Ospedale Ostetrico Ginecologico S. Anna Di Torino - Oncologia Medica, Torino, To
  - Ospedale Mauriziano Umberto I - Ginecologia Oncologica, Torino, TO
  - Ospedale Sacro Cuore - Don Calabria - Oncologia Medica, Negrar, VR

IPD SHARING:
Plan to Share IPD: Undecided